CLINICAL TRIAL: NCT04311541
Title: National, Multicentre, Observational, Non-Interventional Prospective Study of Dexlansoprazole MR in GERD Patients in the Russian Federation
Brief Title: A Study of Dexlansoprazole Modified Release (MR) in Gastroesophageal Reflux Disease (GERD) Participants in the Russian Federation
Acronym: INTEGRO
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision; No Safety Or Efficacy Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MACS-2019-102840; U1111-1247-2413 (Registry Identifier: WHO)
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dexlansoprazole: Participants diagnosed with GERD and initiated treatment with dexlansoprazole MR therapy will be observed prospectively at 150 sites in Russian federation for a period of 2 months.

SUMMARY:
The primary purpose of the study is to evaluate effect of Dexilant treatment among GERD participants in the Russian Federation.

DETAILED DESCRIPTION:
This is an observational, prospective non-interventional study of participants with GERD. This study will evaluate the effect of dexlansoprazole treatment among participants with GERD.

The study will enroll approximately 1500 participants. Due to non-interventional design of the study, the decision about GERD treatment strategy for the participant is taken by attending treating physician. All participants will be enrolled in one observational group: dexlansoprazole.

Prospective data will be collected for a period of 2 months. The frequency of the visits will be assigned by each physician according to their routine practice.

The multi-center trial will be conducted in Russia. The overall duration of study will be approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18 or older years of age by the time of enrolment.
2. Confirmed GERD diagnosis (Non-Erosive Reflux Disease (NERD) or Erosive Reflux Diseases (ERD)) on the base of typical clinical features (symptoms), upper endoscopy within last 12 months prior to inclusion and/or GERDq.
3. Participants diagnosed with GERD less than (<) 3 years prior to study entry, with or without treatment with other GERD medications.
4. Participants without concomitant gastrointestinal (GI) conditions of the gastrointestinal tract and with concomitant GI conditions of the gastrointestinal tract as well as other organ systems concomitant conditions.
5. The physician decides to prescribe Dexilant:

   * as monotherapy or
   * as a part of combined therapy
6. Written informed consent, signed before the participation in the study begins.

Exclusion Criteria:

1. Contraindications for proton-pump inhibitors (PPIs) of respective approved local packaging leaflets.
2. Existence of upper gastrointestinal bleeding.
3. History of surgery on esophagus, stomach or duodenum.
4. Primary esophageal motility disease, achalasia, scleroderma, esophageal / pyloric stricture, primary esophageal spasm, infectious or inflammatory bowel disease, severe malabsorption, severe chronic heart failure, serve cardiovascular disease, renal failure, chronic obstructive pulmonary disease (COPD), asthma, liver cirrhosis.
5. Malignant disease of any kind any system or organ within 5 years, except completely recovered skin cancer.
6. Needs in antibiotics due to severe infection.
7. Alanine transaminase (ALT) or Aspartate aminotransferase (AST) >=Upper limit of normal range*3.
8. Current, previous (within the last one year) or planned (for the next one year) participation in interventional clinical trial.
9. Presenting of mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
10. Any other condition, which on the opinion of the investigator may interfere the participant's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in Russian federation diagnosed with GERD will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline (Visit 1) in GERDq Score on Dexilant Treatment Among GERD Participants at Month 1 (Visit 3) | Baseline (Visit 1), Month 1 (Visit 3)
  GERDq is a self-completed participant questionnaire that is used to assess the frequency of following symptoms: heartburn, regurgitation, stomach pain, nausea, sleep disturbance and use of additional medication due to heartburn/regurgitation. Symptom frequency will be assessed for the week passed using following answers: 0 days, 1 day, 2-3 days, and 4-7 days. Each answer will be assigned a score from 0 to 3 (heartburn, regurgitation, sleep disturbance and use of additional medication due to heartburn/regurgitation) or from 3 to 0 (stomach pain, nausea). Total score will be calculated as a sum of 6 individual scores. GERDq score was calculated as sum of these scores, giving a total score ranging from 0 to 18. When GERDq greater than or equal to (>=)8, the participants could be symptom based diagnosed as GERD. Total score of 0 to 2 points=0 percent (%) likelihood of GERD; 3 to 7 points=50% likelihood of GERD; 8 to 10 points=79% likelihood of GERD; 11 to 18 points=89% likelihood of GERD.

SECONDARY OUTCOMES:
Change From Baseline (Visit 1) in Each of the 6 Questions in GERDq on Dexilant Treatment Among the GERD Participants at Months 1 (Visit 3) and 2 (Visit 4) | Baseline (Visit 1), Month 1 (Visit 3) and Month 2 (Visit 4)
  GERDq is a self-completed participant questionnaire that is used to assess the frequency of following symptoms: heartburn, regurgitation, stomach pain, nausea, sleep disturbance and use of additional medication due to heartburn/regurgitation. Symptom frequency will be assessed for the week passed using following answers: 0 days, 1 day, 2-3 days, and 4-7 days. Each answer will be assigned a score from 0 to 3 (heartburn, regurgitation, sleep disturbance and use of additional medication due to heartburn/regurgitation) or from 3 to 0 (stomach pain, nausea). Total score will be calculated as a sum of 6 individual scores. GERDq score was calculated as sum of these scores, giving a total score ranging from 0 to 18. When GERDq greater than or equal to (>=)8, the participants could be symptom based diagnosed as GERD. Total score of 0 to 2 points=0 percent (%) likelihood of GERD; 3 to 7 points=50% likelihood of GERD; 8 to 10 points=79% likelihood of GERD; 11 to 18 points=89% likelihood of GERD.
Change From Baseline (Visit 1) in GERDq Score on Dexilant Treatment Among GERD Participants at Months 1 (Visit 3) and 2 (Visit 4) | Baseline (Visit 1), Month 1 (Visit 3) and Month 2 (Visit 4)
  GERDq is a self-completed participant questionnaire that is used to assess the frequency of following symptoms: heartburn, regurgitation, stomach pain, nausea, sleep disturbance and use of additional medication due to heartburn/regurgitation. Symptom frequency will be assessed for the week passed using following answers: 0 days, 1 day, 2-3 days, and 4-7 days. Each answer will be assigned a score from 0 to 3 (heartburn, regurgitation, sleep disturbance and use of additional medication due to heartburn/regurgitation) or from 3 to 0 (stomach pain, nausea). Total score will be calculated as a sum of 6 individual scores. GERDq score was calculated as sum of these scores, giving a total score ranging from 0 to 18. When GERDq greater than or equal to (>=)8, the participants could be symptom based diagnosed as GERD. Total score of 0 to 2 points=0 percent (%) likelihood of GERD; 3 to 7 points=50% likelihood of GERD; 8 to 10 points=79% likelihood of GERD; 11 to 18 points=89% likelihood of GERD.
Changes From Baseline (Visit 1) in Daytime Severity GERD Symptoms by Likert Scale on Dexilant Treatment Among GERD Participants at Months 1 (Visit 3) and 2 (Visit 4) | Baseline (Visit 1), Month 1 (Visit 3) and Month 2 (Visit 4)
  Participants collected GERD-associated symptoms of daytime regurgitation, dysphagia, stomach pain, in daily symptom diary. Daytime episodes are defined as those that occurred after arising in the morning until retiring in the evening. The severity score was calculated was based on a 5-point Likert scale ranging from 0 (no symptom) to 4 (very severe symptom); higher scores indicated greater disease activity.
Changes From Baseline (Visit 1) in Nocturnal Severity GERD Symptoms by Likert Scale on Dexilant Treatment Among GERD Participants at Months 1 (Visit 3) and 2 (Visit 4) | Baseline (Visit 1), Month 1 (Visit 3) and Month 2 (Visit 4)
  Participants collected GERD-associated symptoms of night time regurgitation, dysphagia, stomach pain, in daily symptom diary. Night time episodes are defined as those that occurred during the night while sleeping or trying to sleep. The severity score was calculated was based on a 5-point Likert scale ranging from 0 (no symptom) to 4 (very severe symptom); Higher scores indicated greater disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.